CLINICAL TRIAL: NCT04999514
Title: Examining the Effects of Parenting Interventions on Children With Attention-Deficit / Hyperactivity Disorder (AD/HD) and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EA200195
Record Dates: First submitted 2021-07-05; First posted 2021-08-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-07

CONDITIONS: Parenting Intervention; ADHD; Emotion Regulation
Keywords: Mindful parenting; Emotion coaching; Parenting practice; Parenting stress
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: A randomized controlled design will be adopted. There will be two intervention groups, namely Mindful Parenting group and Tuning in to Kids group, and also one waitlist control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not have prior knowledge of the interventions that they will be assigned to.
  The research assistants who support data collection do not know the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful Parenting Program (Experimental): The Mindful Parenting program as developed by Bögels and Restifo (2013), is selected as one of the parenting intervention programs in this study. It is an 8-week program that trains parents in mindfulness and support them to apply mindfulness in parenting context.
  Interventions: Behavioral: Mindful Parenting, Tuning in to Kids
- Tuning in to Kids Program (Experimental): The Tuning in to Kids program as developed by Havighurst and colleagues (2010), is selected as one of the parenting intervention programs in this study. It will be extended to 8-week program that aims at equipping parents with emotion coaching skills.
  Interventions: Behavioral: Mindful Parenting, Tuning in to Kids
- Waitlist Control Group (No Intervention): The waitlist control group will not receive any intervention until the intervention arms complete their training. Depending on the availability of the program instructor, either the Mindful Parenting or Tuning in to Kids program will be offered to this group.

INTERVENTIONS:
Behavioral: Mindful Parenting, Tuning in to Kids — The Mindful Parenting program consists of 8 weekly 2.5-hour group sessions and 3 weekly individual telephone interview sessions (each lasts for around 15-20 minutes). Program materials are translated into Chinese by local partners of the program developer. The Tuning in to Kids program consists of 8 weekly sessions, each lasting for 2.5 hours. Program materials are translated into Chinese.
  Arms: Mindful Parenting Program; Tuning in to Kids Program

SUMMARY:
This study investigates the effects of parenting interventions on improving the emotion regulation and functioning of the children with AD/HD as well as their parents' parenting practices and psychological well-being. Two kinds of parenting interventions are selected in this study, namely the Mindful Parenting and Tuning in to Kids programs. The value of this project lies in empowering parents through parenting techniques which they can use both for themselves and for their daily interactions with children. It is hoped to alleviate their stress from the role of parenting children with special needs, which may in turn lead to their better psychological well-being and greater harmony in the families.

DETAILED DESCRIPTION:
Attention-Deficit / Hyperactivity Disorder (AD/HD) is one of the most common neurodevelopmental disorders affecting children and adolescents. Core symptoms of inattention, hyperactivity and impulsivity are associated with impairments in multiple aspects of functioning. Apart from the cognitive and behavioral symptoms listed in the diagnostic manual, emotional symptoms are often observed by the parents and teachers and commonly reported in behavioral rating scales. The prevalence of emotion-related problems among children and adolescents diagnosed with AD/HD is estimated to be between 24-50%. Emotion regulation problems in children and youths with AD/HD were associated with greater risk for more psychopathology, poorer psychosocial functioning, and increased rate of treatment service utilization. Follow-up study of children with AD/HD into adulthood found a higher prevalence of difficulties in emotion regulation among those with persistent AD/HD symptoms than those without.

Parenting a child with special needs such as AD/HD is known to be associated with increased level of parental stress. Apart from their jobs and other family duties, the parents must meet the challenges of taking care of their children's special needs and dealing with their functional problems. According to a survey conducted by the Centre for Special Educational Needs and Inclusive Education of the Educational University of Hong Kong in 2018, 82% of the parents of children with AD/HD experienced higher level of stress in relation to their children's symptoms, and over half of them reported to have mood problems. The parents often reported great frustrations in bringing up their children with limited support and encountering difficulties in daily interactions with their children. Previous research has demonstrated that parental mental health problems can adversely affect their parenting abilities and their children's adjustment.

Medication and behavioral treatment are the two evidence-based treatments for children with AD/HD. Apart from them, there are programs offered by public hospitals, government departments, and non-governmental organizations on teaching the parents skills to manage behavioral problems of children with AD/HD. However, parents may experience difficulties in applying these behavioral management skills when they are suffering from significant distress. In the recent years, new approaches such as mindfulness and emotion coaching have been applied to parenting intervention programs. Intervention studies have supported that these new parenting approaches have not only brought benefits to the parenting behaviors and parents' mental health but also to the children's behavioral problems and children's psychological well-being. Specific to the emotion regulation of children with AD/HD, the effect of behavioral management parent training has been examined in the previous research. However, there has been very limited intervention study which directly investigates the effect of new parenting intervention approaches on improving the emotion regulation of children.

In the present study, we propose to apply two parenting interventions for improving emotion regulation of children with AD/HD as well as their parents' parenting practices and psychological well-being. The two selected interventions are "Mindful Parenting" program and "Tuning into Kids" program. Using mindfulness techniques and everyday practice, the former intervention aims at helping parents cultivate awareness and self-regulation in parent-child interactions, bring compassion and non-judgmental acceptance to their difficulties. The latter intervention teaches the parents emotion coaching techniques to become more aware and reduce automatic response patterns to their children's emotions, and to communicate understanding of such emotions to children. Research has showed that these two new approaches are related to lower level of parental stress and reactivity, and fewer negative parent-child interactions.

Study Objectives:

1. To evaluate the effects of the two parenting interventions on improving emotion regulation of children with AD/HD as well as their functioning.
2. To evaluate the effects of the two parenting interventions in promoting parents' parenting practices and psychological well-being, which includes their emotion regulation, parenting stress, and mental health conditions.

Hypotheses:

1. It is hypothesized that improvements in emotion regulation and functioning will be observed among children whose parents have completed one of the parenting interventions. Some of the improvements will be sustained in the two-months post-intervention assessment.
2. It is expected that the parents who have completed the one of the parenting interventions will show improvements in their parenting practices and psychological well-being. The improvements will be showed immediately after the intervention, and some of the gains will also be sustained in the two-months post-intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

* The parent who has a child with the diagnosis of AD/HD made by qualified professionals. The child does not have co-morbid developmental disabilities such as Autism Spectrum Disorder and Intellectual Disability.
* The child is attending P.1 to P.4 in local primary schools, age between 6 and 10.

Exclusion Criteria:

* Parent who has previously received training in Mindful Parenting, Tuning in to Kids, or other 8-weeks mindfulness program.
* Parent who has serious mental health condition that rendering him/her incapable of participating in the intervention program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Mindful parenting practice | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]
Mindful parenting practice | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]
Mindful parenting practice | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]
Emotion coaching practice | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Parent Emotional Style Questionnaire (PESQ) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parent emotional style in a particular subscale)]
Emotion coaching practice | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Parent Emotional Style Questionnaire (PESQ) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parent emotional style in a particular subscale)]
Emotion coaching practice | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Parent Emotional Style Questionnaire (PESQ) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parent emotional style in a particular subscale)]
Parents' psychological well-being | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Depression Anxiety Stress Scale 21 (DASS 21) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of depression, anxiety or stress in the respective subscale)]
Parents' psychological well-being | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Depression Anxiety Stress Scale 21 (DASS 21) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of depression, anxiety or stress in the respective subscale)]
Parents' psychological well-being | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Depression Anxiety Stress Scale 21 (DASS 21) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of depression, anxiety or stress in the respective subscale)]
Parenting stress | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Parenting Stress Index - Short Form (PSI-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating higher parental distress or more perceived problems in a particular subscale)]
Parenting stress | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Parenting Stress Index - Short Form (PSI-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating higher parental distress or more perceived problems in a particular subscale)]
Parenting stress | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Parenting Stress Index - Short Form (PSI-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating higher parental distress or more perceived problems in a particular subscale)]
Parents' emotion regulation | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating poorer emotional regulation)]
Parents' emotion regulation | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating poorer emotional regulation)]
Parents' emotion regulation | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating poorer emotional regulation)]
Children's emotion regulation | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Emotion Regulation Index of The Behavior Rating Inventory of Executive Function - Second Edition (BRIEF2) [Min. Value: 1; Max Value: 3 (with higher score indicating more problems in children's emotion regulation)]
Children's emotion regulation | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Emotion Regulation Index of The Behavior Rating Inventory of Executive Function - Second Edition (BRIEF2) [Min. Value: 1; Max Value: 3 (with higher score indicating more problems in children's emotion regulation)]
Children's emotion regulation | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Emotion Regulation Index of The Behavior Rating Inventory of Executive Function - Second Edition (BRIEF2) [Min. Value: 1; Max Value: 3 (with higher score indicating more problems in children's emotion regulation)]

SECONDARY OUTCOMES:
Parent-child relationship | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Parent-child relationship | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Parent-child relationship | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Children's inattention, hyperactivity and impulsivity symptoms | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of inattention or hyperactivity/impulsivity in the respective subscale)]
Children's inattention, hyperactivity and impulsivity symptoms | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of inattention or hyperactivity/impulsivity in the respective subscale)]
Children's inattention, hyperactivity and impulsivity symptoms | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) [Min. Value: 0; Max Value: 3 (with higher score indicating more symptoms of inattention or hyperactivity/impulsivity in the respective subscale)]
Children's functioning | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Strengths and Difficulties Questionnaire (SDQ) [Min. Value: 0; Max Value: 2 (with higher score indicating more child behavioral or social difficulties in a particular subscale)]
Children's functioning | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Strengths and Difficulties Questionnaire (SDQ) [Min. Value: 0; Max Value: 2 (with higher score indicating more child behavioral or social difficulties in a particular subscale)]
Children's functioning | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Strengths and Difficulties Questionnaire (SDQ) [Min. Value: 0; Max Value: 2 (with higher score indicating more child behavioral or social difficulties in a particular subscale)]
General parenting practice | Pre-intervention (within 4 weeks before the commencement of parenting program)
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in a particular subscale)]
General parenting practice | Immediate Post-intervention (within 4 weeks after the completion of parenting program)
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in a particular subscale)]
General parenting practice | Delayed Post-intervention (follow-up 2 months later, waitlist control group not included)
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in a particular subscale)]

CONTACTS AND LOCATIONS:
Overall Officials: Iris Kit Yee LAM, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Background] Anastopoulos, A. D., Smith, T. F., Garrett, M. E., Morrissey-Kane, E., Schatz, N. K., Sommer, J. L., & Ashley-Koch, A. (2011). Self-regulation of emotion, functional impairment, and comorbidity among children with AD/HD. Journal of attention disorders, 15(7), 583-592. Barkley, R. A., & Fischer, M. (2010). The unique contribution of emotional impulsiveness to impairment in major life activities in hyperactive children as adults. Journal of the American Academy of Child & Adolescent Psychiatry, 49(5), 503-513. Beer, M., Ward, L., & Moar, K. (2013). The relationship between mindful parenting and distress in parents of children with an autism spectrum disorder. Mindfulness, 4(2), 102-112. Biederman, J., Spencer, T. J., Petty, C., Hyder, L. L., O'Connor, K. B., Surman, C. B., & Faraone, S. V. (2012). Longitudinal course of deficient emotional self-regulation CBCL profile in youth with ADHD: prospective controlled study. Neuropsychiatric disease and treatment, 8, 267. Bögels, S., Hoogstad, B., van Dun, L., de Schutter, S., & Restifo, K. (2008). Mindfulness training for adolescents with externalizing disorders and their parents. Behavioural and cognitive psychotherapy, 36(2), 193. Bögels, S. M., Hellemans, J., van Deursen, S., Römer, M., & van der Meulen, R. (2014). Mindful parenting in mental health care: effects on parental and child psychopathology, parental stress, parenting, coparenting, and marital functioning. Mindfulness, 5(5), 536-551. Bögels, S. M., Lehtonen, A., & Restifo, K. (2010). Mindful parenting in mental health care. Mindfulness, 1(2), 107-120. Bögels, S., & Restifo, K. (2013). Mindful parenting: A guide for mental health practitioners. Springer Science & Business Media. Gouveia, M. J., Carona, C., Canavarro, M. C., & Moreira, H. (2016). Self-compassion and dispositional mindfulness are associated with parenting styles and parenting stress: The mediating role of mindful parenting. Mindfulness, 7(3), 700-712. Havighurst, S. S., Wilson, K. R., Harley, A. E., Prior, M. R., & Kehoe, C. (2010). Tuning in to Kids: improving emotion socialization practices in parents of preschool children-findings from a community trial. Journal of Child Psychology and Psychiatry, 51(12), 1342-1350. Havighurst, S. S., Wilson, K. R., Harley, A. E., Kehoe, C., Efron, D., & Prior, M. R. (2013). "Tuning into Kids": Reducing young children's behavior problems using an emotion coaching parenting program. Child Psychiatry & Human Development, 44(2), 247-264. Leinonen, J. A., Solantaus, T. S., & Punamäki, R. L. (2003). Parental mental health and children's adjustment: The quality of marital interaction and parenting as mediating factors. Journal of child psychology and psychiatry, 44(2), 227-241. Podolski, C. L., & Nigg, J. T. (2001). Parent stress and coping in relation to child ADHD severity and associated child disruptive behavior problems. Journal of clinical child psychology, 30(4), 503-513. Shaw, P., Stringaris, A., Nigg, J., & Leibenluft, E. (2014). Emotion dysregulation in attention deficit hyperactivity disorder. American Journal of Psychiatry, 171(3), 276-293. Singh, N. N., Lancioni, G. E., Winton, A. S., Singh, J., Singh, A. N., Adkins, A. D., & Wahler, R. G. (2010). Training in mindful caregiving transfers to parent-child interactions. Journal of Child and Family Studies, 19(2), 167-174. Townshend, K., Jordan, Z., Stephenson, M., & Tsey, K. (2016). The effectiveness of mindful parenting programs in promoting parents' and children's wellbeing: a systematic review. JBI database of systematic reviews and implementation reports, 14(3), 139-180. Van der Oord, S., Prins, P. J., Oosterlaan, J., & Emmelkamp, P. M. (2008). Efficacy of methylphenidate, psychosocial treatments and their combination in school-aged children with ADHD: a meta-analysis. Clinical psychology review, 28(5), 783-800. Van der Oord, S., Bögels, S. M., & Peijnenburg, D. (2012). The effectiveness of mindfulness training for children with ADHD and mindful parenting for their parents. Journal of child and family studies, 21(1), 139-147. Webster-Stratton, C. H., Reid, M. J., & Beauchaine, T. (2011). Combining parent and child training for young children with ADHD. Journal of Clinical Child & Adolescent Psychology, 40(2), 191-203. Zhang, D., Chan, S. K. C., Lo, H. H. M., Chan, C. Y. H., Chan, J. C. Y., Ting, K. T., & Wong, S. Y. S. (2017). Mindfulness-based intervention for Chinese children with ADHD and their parents: a pilot mixed-method study. Mindfulness, 8(4), 859-872.